CLINICAL TRIAL: NCT00005234
Title: Cardiovascular Disease in Black Versus White Physicians
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1114; R01HL042734 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2000-04

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Hypertension

SUMMARY:
To examine the natural histories of coronary artery disease and hypertension in cohorts of Black and white men of identical education and occupations.

DETAILED DESCRIPTION:
BACKGROUND:

Prior studies of Black-white differences in hypertension and coronary disease have compared racial groups from markedly different socioeconomic and educational backgrounds. This study represented one of a few, if any, long term prospective studies of cardiovascular disease in middle-class Blacks and whites of similar education and occupation, in whom both youthful and midlife risk factors were assessed.

DESIGN NARRATIVE:

In this prospective study, the prevalence and incidence of coronary artery disease, hypertension, and other cardiovascular diseases were compared using standardized endpoint criteria. The prevalence of cardiovascular risk factors in midlife were compared between cohorts, and included smoking, diabetes, family history, dietary factors, and lipoprotein cholesterol levels. The youthful predictors of midlife cardiovascular risk factors were determined using baseline data collected by identical protocols in the two cohorts between 1957 and 1965. The youthful risk factors were related to the incidence of disease in midlife in two cohorts to identify differences in significance, independence, and relative importance of risk factors in Blacks versus whites.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1988-09; Study Completion 1993-08 (Actual)

REFERENCES:
- [Background] Gelber AC, Klag MJ, Mead LA, Thomas J, Thomas DJ, Pearson TA, Hochberg MC. Gout and risk for subsequent coronary heart disease. The Meharry-Hopkins Study. Arch Intern Med. 1997 Jul 14;157(13):1436-40. PMID 9224221
- [Background] Coresh J, Klag MJ, Mead LA, Liang KY, Whelton PK. Vascular reactivity in young adults and cardiovascular disease. A prospective study. Hypertension. 1992 Feb;19(2 Suppl):II218-23. doi: 10.1161/01.hyp.19.2_suppl.ii218. PMID 1735583
- [Background] Roubenoff R, Klag MJ, Mead LA, Liang KY, Seidler AJ, Hochberg MC. Incidence and risk factors for gout in white men. JAMA. 1991 Dec 4;266(21):3004-7. PMID 1820473
- [Background] Klag MJ, Mead LA, LaCroix AZ, Wang NY, Coresh J, Liang KY, Pearson TA, Levine DM. Coffee intake and coronary heart disease. Ann Epidemiol. 1994 Nov;4(6):425-33. doi: 10.1016/1047-2797(94)90001-9. PMID 7804496
- [Background] Klag MJ, He J, Mead LA, Ford DE, Pearson TA, Levine DM. Validity of physicians' self-reports of cardiovascular disease risk factors. Ann Epidemiol. 1993 Jul;3(4):442-7. doi: 10.1016/1047-2797(93)90074-e. PMID 8275223
- [Background] Klag MJ, Ford DE, Mead LA, He J, Whelton PK, Liang KY, Levine DM. Serum cholesterol in young men and subsequent cardiovascular disease. N Engl J Med. 1993 Feb 4;328(5):313-8. doi: 10.1056/NEJM199302043280504. PMID 8419817